CLINICAL TRIAL: NCT00700206
Title: Phase 2 Randomized Study Comparing Two Dose Schedules of Ezatiostat Hydrochloride (Telintra™, TLK199 Tablets) in Low to Intermediate-1 Risk Myelodysplastic Syndrome (MDS)
Brief Title: Phase 2 Study Comparing Two Dose Schedules of Telintra™ in Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Telik (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLK199.2101
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-08

CONDITIONS: Myelodysplastic Syndrome (MDS)
Keywords: Hematology; MDS; Myelodysplastic Syndrome; Low Risk MDS; Intermediate-1 risk MDS; Int-1 risk MDS; Telintra; ezatiostat hydrochloride; ezatiostat; TLK199; Glutathione; Glutathione analog; Glutathione Transferase; Glutathione Transferase inhibitor; Glutathione Transferase P1-1 inhibitor; GSTp1-1 inhibitor; Apoptosis; Differentiation; Enzyme inhibitor
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — gamma-Glu-S-BzCys-PhGly diethyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Dose Schedule 1: Two weeks treatment with Telintra 3000 mg per day in two divided doses followed by one week with no treatment per three week cycle.
  Interventions: Drug: Ezatiostat Hydrochloride
- 2 (Experimental): Dose Schedule 2: Three weeks treatment with Telintra 2000 mg per day in two divided doses followed by one week with no treatment per four week cycle.
  Interventions: Drug: Ezatiostat Hydrochloride

INTERVENTIONS:
Drug: Ezatiostat Hydrochloride — Dose Schedule 1-3000 mg orally per day in two divided doses for two weeks followed by 1 week with no treatment per three week cycle.
  Dose Schedule 2-2000 mg orally per day in two divided doses for three weeks followed by 1 week with no treatment per four week cycle.
  Other Names: Telintra; ezatiostat tablets

SUMMARY:
This is a randomized, open label, multicenter, Phase 2 study comparing two dose schedules of Telintra in patients with Low or Intermediate-1 risk MDS. Patients at least 18 years of age presenting with histologically confirmed Low to Intermediate-1 risk MDS with documented significant cytopenia for at least two months by the IWG criteria are eligible.

ELIGIBILITY:
Inclusion Criteria:

* Primary or de novo MDS
* Low or intermediate-1 MDS
* ECOG performance status 0 or 1
* Documented significant anemia with or without neutropenia and/or thrombocytopenia
* Adequate kidney and liver function
* Patients must have discontinued hematopoietic growth factors at least 3 weeks prior to study entry

Exclusion Criteria:

* Prior allogenic bone marrow transplant for MDS
* History of MDS IPSS score greater than 1.0
* Pregnant or lactating women
* Any severe concurrent disease, infection, or comorbidity that, in the judgement of the investigator, would make the patient inappropriate for study entry
* Oral steroids e.g. prednisone >10 mg per day
* History of active hepatitis B or C
* Known history of HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Hematologic Improvement-Erythroid (HI-E) rate | 24 Weeks

SECONDARY OUTCOMES:
Hematologic Improvement-Neutrophil (HI-N) rate, the Hematologic Improvement-Platelet (HI-P) rate, overall hematologic response rate, safety profile and Quality of Life assessments. | 24 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gail Brown, MD, Study Director — Telik
Locations (36):
- United States (36):
  - Arizona Cancer Center, Tucson, Arizona
  - Central Hematology Oncology Medical Group, Inc., Alhambra, California
  - St. Jude Heritage Healthcare, Fullerton, California
  - Wilshire Oncology Medical Group, Inc., La Verne, California
  - UCLA Medical Center, Los Angeles, California
  - Clinical Trials and Research Associates, Inc., Montebello, California
  - North Valley Hematology/Oncology Medical Group, Northridge, California
  - Bay Area Cancer Research Group, Pleasant Hill, California
  - Desert Hematology Oncology Medical Group, Rancho Mirage, California
  - Cancer Care Associates Medical Group, Inc., Redondo Beach, California
  - Sansum Clinic, Santa Barbara, California
  - Santa Barbara Hematology Medical Group, Inc., Santa Barbara, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - University of Colorado at Denver Health Sciences Center, Aurora, Colorado
  - The Center for Hematology Oncology, Boca Raton, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northeast Georgia Cancer Care, LLC, Athens, Georgia
  - Suburban Hematology-Oncology Associates, P.C., Lawrenceville, Georgia
  - Joliet Oncology-Hematology Associates, Ltd., Joliet, Illinois
  - Loyola University Chicago, Maywood, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Central Hematology Oncology Medical Group, Inc., Terre Haute, Indiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - St. Vincent's Comprehensive Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Case Western Reserve University/University Hospitals of Cleveland, Cleveland, Ohio
  - Hematology & Medical Oncology, Cleveland, Ohio
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Cancer Care Associates, Tulsa, Oklahoma
  - Kaiser Permanente, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas